CLINICAL TRIAL: NCT02370745
Title: Characterizing the Incretin Effect of Amino Acids (AA) and Defining the Effect of GLP-1 on Muscle Microvascular Blood Flow and Muscle Protein and Glucose Metabolism in Older Age.
Brief Title: Characterizing the Incretin Effect of Amino Acids and Defining GLP-1 Role on Skeletal Muscle
Acronym: Incretin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: G12122013 MSGEM
Record Dates: First submitted 2014-11-10; First posted 2015-02-25 (Estimated); Last update posted 2018-05-02 (Actual); Status verified 2018-03

CONDITIONS: Sarcopenia
Keywords: Incretin; GLP-1; Skeletal muscle metabolism; Microvascular recruitment; Amino Acids; Microvascular blood flow
MeSH Terms: conditions — Sarcopenia | interventions — Glucagon-Like Peptide 1; Incretins; insulin, neutral; Insulin; Amino Acids

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- Post absorptive insulin without GLP-1 (Experimental): Subjects with receive post absorptive insulin concentrations while measures of muscle metabolism and microvascular blood flow are taken through the acute study hours.
  The intervention in this group is Insulin Actrapid to achieve post absorptive insulin levels and glucose infusion to achieve postprandial glucose levels of 7.0-7.5 mmol/L . This will form base line measurement for the next arm which will receive GLP-1 in addition.
  Interventions: Drug: Insulin Actrapid
- Postabsorptive insulin with GLP-1 (Experimental): Subjects will receive post absorptive insulin concentrations with GLP-1 while measures of muscle metabolism and microvascular blood flow are taken through the acute study hours. This arm will cross over with the previous arm.
  The intervention in this group is in the form of GLP-1, Insulin Actrapid to achieve post absorptive insulin levels and glucose infusion to achieve postprandial glucose levels of 7.0-7.5 mmol/L .
  Interventions: Drug: GLP-1; Drug: Insulin Actrapid
- Postprandial insulin without GLP-1 (Experimental): Subjects will receive postprandial insulin concentrations without GLP-1 while measures of muscle metabolism and microvascular blood flow are taken through the acute study hours.
  The intervention in this group is Insulin Actrapid to achieve postprandial insulin levels and glucose infusion to achieve postprandial glucose levels of 7.0-7.5 mmol/L . This will form base line measurement for the next arm which will receive GLP-1 in addition
  Interventions: Drug: Insulin Actrapid
- Postprandial insulin with GLP-1 (Experimental): Subjects with receive postprandial insulin concentrations with GLP-1 while measures of muscle metabolism and microvascular blood flow are taken through the acute study hours. This arm will cross over with the previous arm.
  The intervention in this group is in the form of GLP-1, Insulin Actrapid to achieve postprandial insulin levels and glucose infusion to achieve postprandial glucose levels of 7.0-7.5 mmol/L .
  Interventions: Drug: GLP-1; Drug: Insulin Actrapid
- Oral amino acids-Young (Experimental): Gut hormones will be measured post oral drink containing 15 g of amino acids in young persons. This will cross over with the following 2 arms.
  The intervention here is: 15g of mixed essential amino acid drink.
  Interventions: Dietary Supplement: Oral amino acids
- Intravenous (IV) amino acids- Young (Experimental): Gut hormones will be measured after intravenous amino acid infusion delivering iso equivalent amount of amino acids in young persons.
  The intervention in this group: Intravenous amino acids delivering iso-equivalent amount of 15g mixed essential amino acids
  Interventions: Drug: Intravenous amino acids
- IV amino acids, GLP-1, GIP -Young (Experimental): Gut hormones will be measured after intravenous amino acid infusion delivering iso equivalent amount of amino acids, GLP-1, GIP in young persons.
  The intervention in this group: Intravenous amino acids iso-equivalent to oral 15 g mixed essential amino acids, GLP-1 infusion and GIP infusion
  Interventions: Drug: GLP-1; Drug: GIP; Drug: Intravenous amino acids
- Oral amino acids- Older (Experimental): Gut hormones will be measured post oral drink containing 15 g of mixed essential amino acids in older persons.
  The intervention in this arm: 15 gram of oral mixed essential amino acid drink
  Interventions: Dietary Supplement: Oral amino acids

INTERVENTIONS:
Drug: GLP-1 — GLP-1 effects on skeletal muscle glucose and amino acid metabolism and microvascular blood flow will be scrutinised under the specified insulin concentrations. It will also be used to test the effect of intravenous feed on insulin secretion.
  Other Names: Incretin
  Arms: IV amino acids, GLP-1, GIP -Young; Postabsorptive insulin with GLP-1; Postprandial insulin with GLP-1
Drug: Insulin Actrapid — Skeletal muscle metabolic and microvascular parameters will be tested under specified insulin concentrations with or without GLP-1
  Other Names: Actrapid
  Arms: Post absorptive insulin without GLP-1; Postabsorptive insulin with GLP-1; Postprandial insulin with GLP-1; Postprandial insulin without GLP-1
Dietary Supplement: Oral amino acids — Oral amino acids containing 15 g of amino acids
  Other Names: mixed EAA
  Arms: Oral amino acids- Older; Oral amino acids-Young
Drug: GIP — This will be co infused with GLP-1 and intravenous amino acids
  Other Names: Incretin
  Arms: IV amino acids, GLP-1, GIP -Young
Drug: Intravenous amino acids — This will aim to deliver iso equivalent amount to the amino acids administered orally
  Other Names: IV AA
  Arms: IV amino acids, GLP-1, GIP -Young; Intravenous (IV) amino acids- Young

SUMMARY:
This study has two protocols the aims of which are:

1. To identify age-related effects of AA on incretin secretion and whether and to what extent AA exhibit a true incretin effect (gut- mediated increases in plasma insulin) in younger individuals. (Protocol 1)
2. To define the extra-pancreatic ''novel'', insulin independent effects of glucagon like peptide-1 (GLP-1) on postprandial muscle protein and glucose metabolism and microvascular blood flow. (Protocol 2)

DETAILED DESCRIPTION:
Protocol 1:

This will explore the first aim. 8 Healthy younger volunteers will be recruited to under go 3 arms cross over studies. Interventions will include oral and intravenous amino acids, in addition to intravenous GLP-1 and glucose dependent insulinotropic polypeptide (GIP).

8 older subjects also will be recruited for comparison of the response of GI hormones to amino acids oral feed between young and older men.

Therefore the total number will be recruited to perform this protocol is 16.

Post intervention in all visits, measurements will be taken for:

Insulin, Amino acids, GLP-1, GIP, Ghrelin and peptide YY (PYY).

The measurable end points for this protocol are:

1. Gut hormones levels in response to the 2 methods of AA delivery (I.V and oral)
2. Differences in gut hormones levels between young and older subjects when AA's are delivered orally

Protocol 2:

This will explore the second aim. 16 healthy older subjects will be recruited and subdivided randomly into two groups to receive either post absorptive or postprandial insulin concentrations with or without GLP-1 at physiological ranges in a cross over fashion . During acute study parameters of muscle glucose and amino acids metabolism will be tested together with muscle microvascular recruitment and macro vascular flow in the tested leg.

The measurable end points for this protocol are:

1. Muscle Glucose uptake, assessed by measuring 2-deoxyglucose (2-DOG) phosphate in muscle biopsies
2. Myofibrillar protein synthesis, assessed via muscle biopsy fractional synthesis rate (FSR)
3. Whole Leg Muscle Protein Synthesis, assessed via Arterial-Venous difference (AV method)
4. Whole Leg Muscle Protein Breakdown, assessed via AV method
5. Whole Leg Net Protein Balance, assessed via AV method
6. Muscle microvascular recruitment, assessed via microvascular contrast bubbles filling and refilling post destruction by ultrasound waves.

ELIGIBILITY:
Inclusion Criteria:

- For protocol 1: i. Aged between 18-40 or 65-75 years ii. A body mass index (BMI) >18 and <28 kg/m2

- For Protocol 2: i. Age 65-75 years ii. A body mass index (BMI) >18 and <28 kg/m2

Exclusion Criteria:

* For protocol 1:

  i. A BMI < 18 or > 28 kg·m2 ii. Active cardiovascular disease: uncontrolled hypertension (BP > 160/100), angina, heart failure (class III/IV), arrhythmia, right to left cardiac shunt or recent cardiac event iii. Cerebrovascular disease: previous stroke, aneurysm (large vessel or intracranial) iv. Respiratory disease including pulmonary hypertension, chronic obstructive pulmonary disease (COPD), asthma or an forced expiratory volume in 1 minute (FEV1) less than 1.5 litre.

  v. Metabolic disease: hyper and hypo-parathyroidism, untreated hyper and hypothyroidism, Cushing's disease, types 1 or 2 diabetes vi. Active inflammatory bowel or renal disease vii. Malignancy viii. Recent steroid treatment (within 6 month), or hormone replacement therapy ix. Clotting dysfunction x. Musculoskeletal or neurological disorders xi. Family history of early (<55y) death from cardiovascular disease
* For protocol 2:

Same as protocol 1 in addition to:

i. Overt muscle wasting i.e. muscle mass is more than 1 standard deviation below normal muscle or fat-free mass for age.

ii. Taking beta-adrenergic blocking agents or non-steroidal anti-inflammatory drugs iii. Known sensitivity to SONOVUE or any other drug used in the study. iv. Subject deemed unsuitable for femoral cannulation at screening visit.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Muscle protein and glucose metabolism | 12 months
  Assessed from muscle biopsies taken for measurement of protein synthesis and breakdown and glucose uptake.

SECONDARY OUTCOMES:
Leg Microvascular blood flow | 12 months
  Assessed via contrast enhanced ultrasound.
Leg Macrovascular blood flow | 12 months
  Assessed via ultrasound doppler scans
Insulin secretion in response to oral and intravenous amino acids to assess their ability to exert incretin effect. | 12 months
  Assessed via serial blood draws measuring insulin level at baseline and and post intervention.
Gut hormones secretion in response to amino acids in young and older people | 12 months
  Assessed via serial blood draws measuring gut hormones at baseline and post intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Philip Atherton, PhD, Principal Investigator — University of Nottingham; Iskandar Idris, DM, FRCP, Principal Investigator — University of Nottingham
Locations (1):
- Division of Medical Sciences and Graduate Entry Medicine - School of Medicine - University of Nottingham, Derby, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Nilsson M, Holst JJ, Bjorck IM. Metabolic effects of amino acid mixtures and whey protein in healthy subjects: studies using glucose-equivalent drinks. Am J Clin Nutr. 2007 Apr;85(4):996-1004. doi: 10.1093/ajcn/85.4.996. PMID 17413098
- [Background] Hall WL, Millward DJ, Long SJ, Morgan LM. Casein and whey exert different effects on plasma amino acid profiles, gastrointestinal hormone secretion and appetite. Br J Nutr. 2003 Feb;89(2):239-48. doi: 10.1079/BJN2002760. PMID 12575908
- [Background] Wilkes EA, Selby AL, Atherton PJ, Patel R, Rankin D, Smith K, Rennie MJ. Blunting of insulin inhibition of proteolysis in legs of older subjects may contribute to age-related sarcopenia. Am J Clin Nutr. 2009 Nov;90(5):1343-50. doi: 10.3945/ajcn.2009.27543. Epub 2009 Sep 9. PMID 19740975
- [Background] Sjoberg KA, Holst JJ, Rattigan S, Richter EA, Kiens B. GLP-1 increases microvascular recruitment but not glucose uptake in human and rat skeletal muscle. Am J Physiol Endocrinol Metab. 2014 Feb 15;306(4):E355-62. doi: 10.1152/ajpendo.00283.2013. Epub 2013 Dec 3. PMID 24302010
- [Background] Chai W, Dong Z, Wang N, Wang W, Tao L, Cao W, Liu Z. Glucagon-like peptide 1 recruits microvasculature and increases glucose use in muscle via a nitric oxide-dependent mechanism. Diabetes. 2012 Apr;61(4):888-96. doi: 10.2337/db11-1073. Epub 2012 Feb 22. PMID 22357961
- [Derived] Abdulla H, Phillips B, Wilkinson D, Gates A, Limb M, Jandova T, Bass J, Lewis J, Williams J, Smith K, Idris I, Atherton P. Effects of GLP-1 Infusion Upon Whole-body Glucose Uptake and Skeletal Muscle Perfusion During Fed-state in Older Men. J Clin Endocrinol Metab. 2023 Mar 10;108(4):971-978. doi: 10.1210/clinem/dgac613. PMID 36260533